CLINICAL TRIAL: NCT04588090
Title: A Prospective Randomized Controlled Study of Radiotherapy and the Concurrent Three-week and Single-week TP Chemotherapy for Advanced Cervical Squamous Cell Carcinoma and the Correlation Between HPV Classification and Sensitivity.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dongling Zou, Director, Chongqing University Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG0105
Record Dates: First submitted 2020-09-30; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — TP protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The concurrent 3 weeks treatment group（external radiation plus intraluminal after-loading irradiation+concurrent platinum-containing 3 weeks chemotherapy）
  Interventions: Procedure: The concurrent 3 weeks TP regimen; Radiation: External radiation plus intraluminal after-loading irradiation
- Standard chemoradiation group (Placebo Comparator): Standard chemoradiation（external radiation plus intraluminal after-loading irradiation+concurrent platinum-containing weekly chemotherapy）
  Interventions: Procedure: The concurrent weekly TP regimen; Radiation: External radiation plus intraluminal after-loading irradiation

INTERVENTIONS:
Procedure: The concurrent 3 weeks TP regimen — paclitaxel + cisplatin regimen (TP-TAX: 150mg/m^2, DDP: 70mg/m^2 (35mg/m^2, d1, d2), 1 time/3 weeks) chemotherapy for 2 cycles.
  Arms: Experimental group
Procedure: The concurrent weekly TP regimen — paclitaxel + cisplatin regimen (TP regimen: TAX 50mg/m^2, DDP: 25mg/m^2) 6 cycles of chemotherapy
  Arms: Standard chemoradiation group
Radiation: External radiation plus intraluminal after-loading irradiation — External radiotherapy of linear accelerator, CT simulation positioning, and intensity modulated radiotherapy will be applied for external radiotherapy. The prescribed dose is 95% PTV 45-50.8Gy/25-28 times (1.8Gy/time), the maximum and minimum in the target area do not exceed ±10% of the prescribed dose, and the increase in enlarged lymph nodes will reach 50-66GY. At the same time, the total dose of 192Ir high-dose rate intraluminal after-loading irradiation is 30-36Gy (EQD2: 40-48GY), and external pelvic irradiation is not available on the day of intraluminal after-loading irradiation.

SUMMARY:
the main purpose for this experiments are as follows: 1. Patients with stage ⅡB-ⅢB cervical squamous cell carcinoma who received full dose radiotherapy will be randomly assigned to the combined TP regimen weekly treatment group and 3-week treatment group for the short-term efficacy and safety observation; 2. All enrolled patients will be tested for HPV subtype infection; the relationship between the sensitivity and curative effect of concurrent radiotherapy and chemotherapy will be analyzed, and at the end of the test, HPV subtypes will be tested again and changes will be analyzed to provide more clinical evidence for the reasonable comprehensive treatment and precision medical treatment of advanced cervical squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. The patient participated in this study voluntarily and all volunteers will sign the informed consent.
2. New cervical squamous cell carcinoma cases between 18 and 70 years old;
3. Clinical stages: stage ⅡB-stage ⅢB;
4. PS score is less than 2 points;
5. Expected survival is over 3 months;
6. Blood routine: Hb≥70g/L, WBC≥3.5×10^9/L, ANC≥1.5×10^9/L, PLT≥80×10^9/L
7. Serum ALT and AST≤2×ULN; serum creatinine≤1.5×ULN;
8. Women of childbearing age must undergo a pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative, and are willing to use appropriate methods of contraception during the trial;
9. Patients who can comply with the trial protocol (judged by the investigator).

Exclusion Criteria:

1. Active or uncontrolled serious infection;
2. Liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral treatments;
3. A history of immunodeficiency, including HIV positive or other acquired congenital immunodeficiency diseases;
4. Chronic renal insufficiency and renal failure;
5. Pregnant woman;
6. Myocardial infarction, severe arrhythmia and congestive heart failure ≥2 (New York Heart Association (NYHA) classification);
7. Patients receiving targeted therapy and pelvic artery embolism;
8. Those who have had arterial/venous thrombosis within 6 months, such as cerebrovascular accident, deep vein thrombosis and pulmonary embolism;
9. Those who have received radiotherapy for malignant pelvic tumors in the past;
10. Patients with autoimmune system diseases such as systemic lupus erythematosus;
11. Patients with comorbidities who need to take drugs with severe liver and kidney damage during treatment, such as tuberculosis;
12. Patients who cannot understand the content of the experiment and cannot cooperate, and those who refuse to sign the informed consent;
13. Those with concomitant diseases or other special circumstances that seriously endanger the safety of patients or affect the completion of the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
disease control rate (DCR) | 1 month and 3 months
  Including the percentage of patients with complete remission, partial remission or with stable disease state and maintained for more than 4 weeks among the patients with evaluable efficacy.
Objective response rate (ORR) | 1 month and 3 months
  Including the percentage of patients with complete remission or partial remission and maintained for more than 4 weeks among the patients with evaluable efficacy.

SECONDARY OUTCOMES:
progression-free survival (PFS) | 2 years
  the time from patient randomization to objective progression or death.
overall survival (OS) | 3 years
  the time from the beginning of enrollment to death for any reason. For subjects who are lost to follow-up, the time of last follow-up is usually calculated as the time of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No